CLINICAL TRIAL: NCT04722081
Title: Virtual Reality Training Combined With a Physical Therapy Program in the Rehabilitation of Patients After Tibial Eminence Fractures
Brief Title: Virtual Reality for Tibial Eminence Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Nehad Ahmed Youness Abo-zaid, Lecturer of physical therapy, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIBIAL EMINENCE
Record Dates: First submitted 2021-01-14; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Tibial Fractures
Keywords: Tibial eminence fracture; Virtual reality
MeSH Terms: conditions — Tibial Fractures; Knee Fractures | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): children received selected physical therapy exercises
  Interventions: Other: physical therapy
- Study Group (Experimental): children received selected physical therapy exercises plus virtual reality training
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: physical therapy — physical therapy-specific exercises

SUMMARY:
Tibial eminence fracture, a bony avulsion of the anterior cruciate ligament (ACL) from its insertion on the intercondylar eminence,1 was first described by Poncet in 1875. 2 Also known as tibial spine fractures, these injuries occur most commonly in skeletally immature patients between the ages of 8 and 14 years

ELIGIBILITY:
Inclusion Criteria:

* age of children from five to nine
* children have fracture in tibial eminence

Exclusion Criteria:

* children have fracture in tibial eminence grade III

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | pain assessment at day 0
  assessment severity of pain
Visual analogue scale | pain assessment at day 180
  assessment severity of pain

SECONDARY OUTCOMES:
A universal goniometer | assessment te range of knee extension at date 0
  assessment te range of knee extension
A universal goniometer | assessment te range of knee extension at date 180
  assessment te range of knee extension

OTHER OUTCOMES:
Pediatric Balance Scale | assessment of balance at date 0
  assessment of balance
Pediatric Balance Scale | assessment of balance at date 180
  assessment of balance

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A Abo-zaid, lecturer, Principal Investigator — South Valley University, Faculty of Physical Therapy
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young W, Ferguson S, Brault S, Craig C. Assessing and training standing balance in older adults: a novel approach using the 'Nintendo Wii' Balance Board. Gait Posture. 2011 Feb;33(2):303-5. doi: 10.1016/j.gaitpost.2010.10.089. Epub 2010 Nov 18. PMID 21087865
- [Background] Wilfinger C, Castellani C, Raith J, Pilhatsch A, Hollwarth ME, Weinberg AM. Nonoperative treatment of tibial spine fractures in children-38 patients with a minimum follow-up of 1 year. J Orthop Trauma. 2009 Aug;23(7):519-24. doi: 10.1097/BOT.0b013e3181a13fe4. PMID 19633462
- [Background] Vander Have KL, Ganley TJ, Kocher MS, Price CT, Herrera-Soto JA. Arthrofibrosis after surgical fixation of tibial eminence fractures in children and adolescents. Am J Sports Med. 2010 Feb;38(2):298-301. doi: 10.1177/0363546509348001. Epub 2009 Dec 23. PMID 20032285